CLINICAL TRIAL: NCT01225081
Title: A Phase III Study to Assess the Efficacy, Safety and Tolerability of ASP1941 in Combination With Pioglitazone in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Pioglitazone Alone
Brief Title: A Study to Assess the Efficacy and Safety of ASP1941 in Combination With Pioglitazone in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1941-CL-0107
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: ASP1941; Diabetes mellitus; pioglitazone
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — ipragliflozin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP group (Experimental): ASP1941 and pioglitazone
  Interventions: Drug: ipragliflozin; Drug: Pioglitazone
- Placebo group (Placebo Comparator): placebo and pioglitazone
  Interventions: Drug: Placebo; Drug: Pioglitazone

INTERVENTIONS:
Drug: ipragliflozin — oral
  Other Names: ASP1941
  Arms: ASP group
Drug: Placebo — oral
  Arms: Placebo group
Drug: Pioglitazone — oral
  Other Names: Actos

SUMMARY:
This study is to evaluate the efficacy and safety after concomitant administration of ASP1941 and pioglitazone in patients with diabetes mellitus.

DETAILED DESCRIPTION:
This study is to evaluate the efficacy (HbA1c change from baseline) and safety of ASP1941 in combination with pioglitazone in subjects with type 2 diabetes mellitus (T2DM) who have inadequate glycemic control with pioglitazone alone. The effects of ASP1941 are compared with those of placebo. Double blind period continues for 24 weeks followed by open period in each patient.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients receiving pioglitazone mono-therapy for at least 4 weeks
* HbA1c value between 7.0 and 9.5%
* Body Mass Index (BMI) 20.0 - 45.0 kg/m2

Exclusion Criteria:

* Type 1 diabetes mellitus patients
* Serum creatinine > upper limit of normal
* Proteinuria (albumin/creatinine ratio > 300mg/g)
* Dysuria and/or urinary tract infection, genital infection
* Significant renal, hepatic or cardiovascular diseases
* Severe gastrointestinal diseases
* Heart failure patients

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2010-09-15 (Actual); Primary Completion 2012-04-28 (Actual); Study Completion 2012-04-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | Baseline and for 24 weeks

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose | Baseline and for 24 weeks
Change from baseline in fasting serum insulin | Baseline and for 24 weeks
Safety as reflected by adverse events, routine safety laboratories, vital signs, physical examinations and 12-lead electrocardiograms (ECGs) | For 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (7):
- Japan (7):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyushu
  - Tōhoku

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Kashiwagi A, Shestakova MV, Ito Y, Noguchi M, Wilpshaar W, Yoshida S, Wilding JPH. Safety of Ipragliflozin in Patients with Type 2 Diabetes Mellitus: Pooled Analysis of Phase II/III/IV Clinical Trials. Diabetes Ther. 2019 Dec;10(6):2201-2217. doi: 10.1007/s13300-019-00699-8. Epub 2019 Oct 12. PMID 31606880
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=101